CLINICAL TRIAL: NCT04669535
Title: A Two-Stage, Dose-Escalation and Safety & Efficacy Study of Bilateral Intraparenchymal Thalamic and Intracisternal/Intrathecal Administration of AXO-AAV-GM2 in Tay-Sachs or Sandhoff Disease
Brief Title: A Dose-escalation and Safety & Efficacy Study of AXO-AAV-GM2 in Tay-Sachs or Sandhoff Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew from the study and there was a lack of funding to complete stage 2 of the designed study.
Sponsor: Terence Flotte (Other)
Collaborators: University of Massachusetts, Worcester (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Terence Flotte, Dean, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXO-GM2-001
Record Dates: First submitted 2020-11-23; First posted 2020-12-17 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Tay-Sachs Disease; Sandhoff Disease
Keywords: GM2 Gangliosidosis; Hexosaminidase A Deficiency; HexA Deficiency; TSD; SD; Lysosomal Storage Disorders; Tay-Sachs Disease; Sandhoff Disease
MeSH Terms: conditions — Tay-Sachs Disease; Sandhoff Disease; Gangliosidoses, GM2; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AXO-AAV-GM2 (Experimental): AXO-AAV-GM2 infusion
  Interventions: Biological: AXO-AAV-GM2 Starting Dose; Biological: AXO-AAV-GM2 Low Dose; Biological: AXO-AAV-GM2 Middle Dose; Biological: AXO-AAV-GM2 High Dose

INTERVENTIONS:
Biological: AXO-AAV-GM2 Starting Dose — 1:1 ratio of AAVrh8-HEXA and AAVrh8-HEXB, administered via bilateral thalamic (BiTh) and dual intracisterna magna (ICM)/intrathecal (IT) administration into the cerebrospinal fluid (CSF).
  Other Names: AAVrh8-HEXA and AAVrh8-HEXB
Biological: AXO-AAV-GM2 Low Dose — 1:1 ratio of AAVrh8-HEXA and AAVrh8-HEXB, administered via bilateral thalamic (BiTh) and dual intracisterna magna (ICM)/intrathecal (IT) administration into the cerebrospinal fluid (CSF).
  Other Names: AAVrh8-HEXA and AAVrh8-HEXB
Biological: AXO-AAV-GM2 Middle Dose — 1:1 ratio of AAVrh8-HEXA and AAVrh8-HEXB, administered via bilateral thalamic (BiTh) and dual intracisterna magna (ICM)/intrathecal (IT) administration into the cerebrospinal fluid (CSF).
  Other Names: AAVrh8-HEXA and AAVrh8-HEXB
Biological: AXO-AAV-GM2 High Dose — 1:1 ratio of AAVrh8-HEXA and AAVrh8-HEXB, administered via bilateral thalamic (BiTh) and dual intracisterna magna (ICM)/intrathecal (IT) administration into the cerebrospinal fluid (CSF).
  Other Names: AAVrh8-HEXA and AAVrh8-HEXB

SUMMARY:
The AXO-GM2-001 study is an open-label, two-stage clinical trial designed to evaluate safety and dose-escalation (Stage 1) and safety and efficacy (Stage 2) of a bilateral thalamic and intracisternal/intrathecal infusion of AXO-AAV-GM2 in pediatric participants with GM2 Gangliosidosis (also known as Tay-Sachs or Sandhoff Diseases), a set of rare and fatal pediatric neurodegenerative genetic disorders caused by defects in the HEXA (leading to Tay-Sachs disease) or HEXB (leading to Sandhoff disease) genes that encode the two subunits of the β-hexosaminidase A (HexA) enzyme. AXO-AAV-GM2 is an investigational gene therapy that aims to restore HexA function by introducing a functional copy of the HEXA and HEXB genes via co-administration of two vectors utilizing the neurotropic adeno-associated virus recombinant human 8 serotype (AAVrh.8) capsid carrying the human HEXA or HEXB cDNA.

The trial is expected to enroll pediatric participants with Tay-Sachs or Sandhoff Diseases, where infantile-onset participants will range from 6 months to 20 months old, and juvenile-onset participants will range from 2 years to 12 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with genetically diagnosed TSD or SD mutations of either HEXA gene or HEXB gene

   a. Stage 1 juvenile-onset participants must be ≥ 2 years old and ≤ 12 years old at time of gene transfer i. Diagnosis consistent with juvenile-onset TSD or SD b. Stage 1 infantile-onset participants must be between 6-20 months of age at the time of gene transfer i. Diagnosis consistent with infantile-onset TSD or SD
2. Juvenile onset participants must demonstrate a minimum of 2 of the following age-appropriate clinical features/abilities, confirmed by the site examiner at the time of screening and reaffirmed prior to the initiation of immunosuppression:

   1. A Gross Motor Function Classification-MLD (GMFC-MLD) score of 0, 1 or 2. The minimum gross motor function (GMFC-MLD level 2) is the 'ability to walk with support and walking without support is not possible (fewer than 5 steps)'. (Participants aged 2-12 years) Note: Any form of support is permitted; however, the participant must initiate each step and complete it for a total of 5 steps.
   2. Fine Motor Function

      * For Participants aged 4-12 years: A Manual Ability Classification System (MACS) score of I, II, III, or IV. The minimum level of manual ability (level IV) corresponds to 'Handles a limited selection of easily managed objects in adapted situations'.
      * For participants aged 2-4 years: attainment of fine motor function/coordination abilities and milestones with normal or a reduced quality of performance. That is, the ability to coordinate fingers and both hands to play, such as swinging a bat or opening a container (pathways.org) OR the ability to use fingertips to pick up small objects, i.e., the child uses pad of his/her thumb and any fingertip to grasp a pellet or small object as described in BSID III Fine Motor Sub-test Item #26. .
   3. Speech:

      * For participants aged 4-12 years, a speech disturbance score of 0, 1, 2 or 3 on the speech disturbance subset of the Scale for Assessment and Rating of Ataxia (SARA). The minimum speech requirement is a speech disturbance in which most words can be understood, with occasional words difficult to understand secondary to dysarthria.
      * Participants aged 2-4 years who have attained the communication milestone of ability to consistently use 2-3 word phrases may be assessed in line with this criterion using the speech disturbance subset of the SARA.
      * For participants aged 2-4 years who have not yet attained the above communication milestone, the minimum requirement is the ability to imitate at least one word, even if the imitation consists of vowels only (BSID III, expressive communication subtest, item #16)
3. Infantile onset participants must demonstrate current* or historical† ability to sit without support for at least 5 seconds

   * As assessed in item 22 of the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) Gross Motor Scale or documented medical records

   † Documented within available medical records

   In addition, infantile onset participants must demonstrate a minimum of 3 of the following developmental skills confirmed by the site examiner at the time of screening and reaffirmed prior to the initiation of immunosuppression:
   1. Head control - While supine, with head in midline turns head symmetrically (score of 3 on GMFM item 1)
   2. Uses hands to support self while sitting
   3. Reach for an object that is held out for them above their chest while supine
   4. Transfer of object from hand to hand while supine
   5. Eye tracking while supine
   6. Looks at an object of interest for at least 3 continuous seconds
4. Surgical readiness for gene transfer by the routes of administration confirmed by the study neurosurgeon*, based on examination and MRI findings

   The following findings will disallow the performance of the BiTh procedure thereby excluding the participant from participation:
   * Any scalp and skull related lesion (e.g., vascular, infectious) over the surgical entry area
   * Any intracranial lesion (e.g., vascular, cystic, other mass lesions), significant immaturity or deformity of the brain anatomy that would make the intended surgical trajectory high risk

   The following findings will disallow the performance of the ICM/IT procedure thereby excluding the participant from participation:
   * Any skin related lesion (e.g., vascular, infectious) over the lumbar puncture site
   * Any intraspinal or intracranial lesion in posterior fossa (e.g., vascular, cystic, other mass lesions) or significantly deformed, distorted brain, spinal and cisternal anatomy that make the intended intrathecal trajectory high risk or not feasible * Participants otherwise eligible for study participation but deemed not currently fit for neurosurgery may be re-screened at the discretion of the investigator
5. Participants receiving off-label Zavesca® (miglustat) and/or Tanganil® (acetyl-leucine) must be willing to discontinue these therapies 30 days prior to the start of screening
6. Ability to reliably travel to the study sites for study visits according to the Schedule of Assessments

Exclusion Criteria:

1. Presence of G269S or W474C mutation in HEXA
2. Evidence of lower respiratory tract aspiration not easily manageable with thickening of feedings or substitution of a modified bottle nipple, as judged on a multi-texture contrast swallow.
3. History of multiple aspiration pneumonias occurring in the past twelve months.
4. Respiratory support in the form of ventilation (invasive or non-invasive).
5. History of drug-resistant seizures or status epilepticus
6. History and/or findings of spinal cord disease that would preclude the lumbar puncture and ICM/IT infusion procedures including:

   * Infectious process involving the spinal canal which may cause adhesions or septations in the spinal and/or subarachnoid space
   * Previous spinal surgeries
   * History of trauma, bleeding in the spinal canal
   * Vascular or cystic lesions, or any other mass lesion
   * Congenital deformities and malformations involving the spinal canal
   * Posterior fossa findings (low lying cerebellar tonsils, crowded foramen magnum, small or absent cisterna manga)
7. The participant's parent(s) or legal guardian(s) is unable to understand the nature, scope, and possible consequences of the study, or does not agree to comply with the protocol-defined schedule of assessments
8. Any prior participation in a study in which a gene therapy vector or stem cell transplantation was administered
9. Immunizations of any kind in the month prior to screening
10. Cardiomyopathy or other cardiac disease based on echocardiogram and/or electrocardiogram, (ECG) that in the opinion of the Investigator would deem the participant unsafe to undergo surgical gene transfer
11. Indwelling ferromagnetic devices that would preclude MRI//MRS/DTI imaging
12. Ongoing medical condition that is deemed by the Investigator to interfere with the conduct or assessments of the study
13. Current clinically significant infections including any requiring systemic treatment including but not limited to human immunodeficiency virus (HIV), Hepatitis A, B, or C
14. History of or current chemotherapy, radiotherapy or other immunosuppressive therapy within the past 30 days. Corticosteroid treatment may be permitted at the discretion of the PI
15. Clinically significant laboratory abnormalities:

    Based on age-specific reference range and determined by the investigator:
    * Total WBC count
    * Hemoglobin
    * Creatinine
    * Pancreatic enzymes

    Based on the following thresholds:
    * Platelet count (< 150,000/μL)
    * Prothrombin (PT), partial thromboplastin time (PTT) >2X normal
    * Liver transaminases (Hy's Law: > 3x elevations above the ULN of ALT or AST and serum total bilirubin > 2xULN)
16. Participants for whom any of the proposed study procedures or medications (i.e., sirolimus, trimethoprim/sulfamethoxazole) would be contraindicated
17. Failure to thrive, defined as falling 20 percentiles (20/100) in body weight in the 3 months preceding Screening/Baseline
18. Participant is not suitable for participation in the study in the opinion of the Principal Investigator

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Flotte, MD, Principal Investigator — University of Massachusetts Medical Health Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Center for Rare Neurological Diseases, Boston, Massachusetts
  - University of Massachusetts Medical Health Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eichler F, Cataltepe OI, Daci R, Puri AS, Taghian T, Jiang X, Shazeeb MS, Kuhn A, Hader A, Celik H, Vardar Z, Lewis CJ, Artinian R, Nagy A, Vachha B, Thompson R, Gallagher T, Bateman S, Parzych J, Spanakis SG, Vaughn TA, Pier K, De Boever E, Abbott MA, D Ambrosio E, Kokoski D, Blackwood M, Drummond E, Ratai EM, Townsend EL, McLaughlin H, Tifft CJ, Keeler AM, Sena-Esteves M, Gray-Edwards HL, Flotte TR. Dual-vector rAAVrh8 gene therapy for GM2 gangliosidosis: a phase 1/2 trial. Nat Med. 2025 Sep;31(9):2927-2935. doi: 10.1038/s41591-025-03822-4. Epub 2025 Aug 15. PMID 40817303
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a dose-escalation study in children affected with GM2 gangliosidosis who were treated in four cohorts at dosage levels ranging from 1.42E+14 to 3.56E+14 vg per patient. All subjects are treated with a 1:1 ratio of AAVrh8-HEXA and AAVrh8-HEXB, administered via bilateral thalamic (BiTh) and dual intracisterna magna (ICM)/intrathecal (IT) administration into the cerebrospinal fluid (CSF). The BiTh injection volume and vector dose was doubled between each cohort.
Pre-assignment Details: The study was initially designed as a 2-stage study with dose escalation in stage 1 and safety and efficacy in stage 2, with the optimal dose identified in stage 1 however due to lack of funding only stage 1 was completed in this study. No subjects were enrolled in stage 2.
Groups:
- AXO-AAV-GM2 Starting Dose: Subjects treated with AXO-AAV-GM2 Starting Dose infusion
- AXO-AAV-GM2 Low Dose: Subjects treated with AXO-AAV-GM2 Low Dose infusion
- AXO-AAV-Middle Dose: Subjects treated with AXO-AAV-GM2 Middle Dose infusion
- AXO-AAV-GM2 High Dose: Subjects treated with AXO-AAV-GM2 High Dose infusion
Period: Overall Study
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-Middle Dose | AXO-AAV-GM2 High Dose
Started | 1 | 3 | 3 | 2
Completed | 0 | 2 | 3 | 2
Not Completed | 1 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects treated with AXO-AAV-GM2
Groups:
- AXO-AAV-GM2 Middle Dose: Subjects treated with AXO-AAV-GM2 Mid Dose Infusion
- Total: Total of all reporting groups
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose | Total
Number analyzed (Participants) | 1 | 3 | 3 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 3 | 2 | 9
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 2 | 8
  Male | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Disease Condition [Count of Participants; unit: Participants]
  Tay-Sachs Disease (Hex A mutation) | 0 | 3 | 2 | 2 | 7
  Sandhoff Disease (Hex B mutation) | 1 | 0 | 1 | 0 | 2
Disease Type [Count of Participants; unit: Participants]
  Infantile Onset | 1 | 1 | 2 | 2 | 6
  Juvenile Onset | 0 | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence, Severity, Seriousness and Relatedness to Treatment of Treatment Emergent Adverse Events
Description: The measure of total numbers of total treatment emergent adverse events (TEAEs), serious adverse events (SAEs) after treatment with the vector whether related or unrelated to treatment as well as the number of adverse events (AEs) related to AXO-AAV-GM2 vector and neurosurgical procedures.
Time Frame: At least through 24 weeks post-treatment (infantile-onset participants) to 48 weeks post-treatment (juvenile-onset participants). All AEs are reported through the transition of the study to long-term follow-up.
Population: All subjects treated with AXO-AAV-GM2 at all doses
Measure: Number; unit: number of events
Groups:
- AXO-AAV-GM2 Starting Dose: Subjects treated with AXO-AAV-GM2 Starting Dose
- AXO-AAV-GM2 Low Dose: Subjects treated with AXO-AAV-GM2 Low Dose
- AXO-AAV-GM2 Middle Dose: Subjects treated with AXO-AAV-GM2 Middle Dose
- AXO-AAV-GM2 High Dose: Subjects treated with AXO-AAV-GM2 High Dose
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
Number analyzed (Participants) | 1 | 3 | 3 | 2
number of events
  Total number of TEAEs | 21 | 43 | 51 | 18
  Total Number of Treatment Emergent SAEs | 1 | 9 | 8 | 1
  AEs Related to Vector | 0 | 4 | 6 | 5
  AEs Related to Neurosurgery | 2 | 4 | 4 | 6

2. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs Per Investigator Assessment
Description: Any abnormal vital signs that the investigator determined was clinically significant was recorded as an adverse event.
Time Frame: 24 weeks (infantile-onset participants) to 48 weeks (juvenile-onset participants)
Measure: Count of Participants; unit: Participants
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
Number analyzed (Participants) | 1 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Physical Exam Per Investigator Assessment
Description: Physical exam findings that the investigator determined to be clinically significant and related to the treatment with AXO-AAV-GM2, surgical procedure or immune suppression.
Time Frame: 24 weeks (infantile-onset participants) to 48 weeks (juvenile-onset participants)
Measure: Count of Participants; unit: Participants
Groups:
- AXO-AAV-GM2 Starting Dose: All subjects treated with AXO-AAV-GM2 Starting Dose
- AXO-AAV-GM2 Low Dose: All subjects treated with AXO-AAV-GM2 Low Dose
- AXO-AAV-GM2 Middle Dose: All subjects treated with AXO-AAV-GM2 Middle Dose
- AXO-AAV-GM2 High Dose: All subjects treated with AXO-AAV-GM2 High Dose
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
Number analyzed (Participants) | 1 | 3 | 3 | 2
Participants
  Dystonia | 0 | 1 | 1 | 0
  Mucositis | 0 | 2 | 2 | 0
  Surgical Site Swelling | 0 | 0 | 1 | 0
  Surgical Wound Drainage | 0 | 0 | 1 | 1
  Wound Dehiscence | 0 | 1 | 1 | 0
  Oral Candidiasis | 1 | 0 | 2 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Clinical Safety Laboratory Tests on Blood/Urine/CSF
Description: Abnormal laboratory findings in subjects treated with AXO-AAV-GM2 that were felt to be clinically significant and reported as adverse events.
Time Frame: 24 weeks (infantile-onset participants) to 48 weeks (juvenile-onset participants)
Population: Subjects treated with AXO-AAV-GM2
Measure: Count of Participants; unit: Participants
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
Number analyzed (Participants) | 1 | 3 | 3 | 2
Participants
  Abnormal results of liver function studies | 0 | 1 | 2 | 2
  Anemia | 1 | 1 | 1 | 1
  Hypokalemia | 0 | 0 | 1 | 1
  Neutropenia | 1 | 0 | 0 | 0

5. Secondary Outcome: Serum Cellular and Antibody Immune Response to Vector Capsid/Transgene
Description: Subjects with clinically significant serum cellular and antibody immune response to vector capsid/transgene that were reported as adverse events and treated with an increase in steroids.
Time Frame: 24 weeks (infantile-onset participants) to 48 weeks (juvenile-onset participants)
Population: Subjects with clinically significant serum cellular and antibody immune response to vector capsid/transgene
Measure: Count of Participants; unit: Participants
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
Number analyzed (Participants) | 1 | 3 | 3 | 2
Participants | 0 | 1 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were captured from screening prior to treatment until the subjects were all moved to long-term follow-up and the initial study was closed. This time ranged from 9 months for the most recently treated patient to 3 years for the patient who was the furthest from their treatment date at the time of moving to long-term follow-up.
Arm/Group | AXO-AAV-GM2 Starting Dose | AXO-AAV-GM2 Low Dose | AXO-AAV-GM2 Middle Dose | AXO-AAV-GM2 High Dose
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXO-AAV-GM2 Starting Dose (N=1) | AXO-AAV-GM2 Low Dose (N=3) | AXO-AAV-GM2 Middle Dose (N=3) | AXO-AAV-GM2 High Dose (N=2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pre-treatment SAE
Wound dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspiration pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Fatal SAE
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza A (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Death due to disease progression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Fatal SAE
Mental status changes (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXO-AAV-GM2 Starting Dose (N=1) | AXO-AAV-GM2 Low Dose (N=3) | AXO-AAV-GM2 Middle Dose (N=3) | AXO-AAV-GM2 High Dose (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutrophil Count Decrease (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coffee Ground Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Reflux (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Rigors (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery-related Pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Surgical Site Swelling (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical Wound Drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound Dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal Results of Liver Function Studies (Hepatobiliary disorders) | 0 (0) | 1 (2) | 2 (3) | 2 (2)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anti-Capsid immune response by ELISpot (Immune system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Seasonal Allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
G-Tube Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pediculosis Capitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Vaginal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PICC Line Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal Movements (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delayed recovery from anesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — These 2 events of dystonia were reported as Adverse Events of Special Interest (AESI)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macrocephaly (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Tardive dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventriculomegaly (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersalivation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Increased Mucus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis due to adhesive (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Seborrheic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision Site Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scalp Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perioral Cyanosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature Ventricular Contractions (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pre-treatment adverse event
Run of Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pre-treatment adverse event
Hiccups (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pre-treatment adverse event
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Pre-treatment adverse event
Procedure-related pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Pre-treatment adverse event
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pre-treatment adverse event
Covid-19 Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pre-treatment adverse event
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Pre-treatment adverse event
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pre-treatment adverse event
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pre-treatment adverse event
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pre-treatment adverse event
Infusion Related Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) — Pre-treatment adverse event

LIMITATIONS AND CAVEATS:
While encouraging, the results of this study also demonstrate important limitations of this therapeutic approach. First, the infusion of 1.25 ml of vector material into the parenchyma of the thalamus likely is at or near the maximum feasible dose. With less than complete clinical efficacy and limited ability to increase the dose further, the clinical utility of this approach is far from optimal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04669535/Prot_SAP_000.pdf